CLINICAL TRIAL: NCT01239706
Title: A Phase IIa, Single Centre, Open Label Study to Characterize the Safety of Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Traumatic Brain Injury: Dosing Tier 1
Brief Title: Safety Study of Human Chorionic Gonadotropin (hCG) and Epoetin Alfa (EPO) in Traumatic Brain Injury: Dosing Tier 1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Stem Cell Therapeutics Corp. (Industry)
Responsible Party: Dr. David A Zygun, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23036
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Epoetin Alfa; Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NTx 265 (Experimental)
  Interventions: Drug: NTx 265

INTERVENTIONS:
Drug: NTx 265 — 10,000IU of hCG, every other day for three doses followed by 4000IU once daily for three days of erythropoietin
  Other Names: Eprex, Ortho Biotech; Ovidrel, Serono

SUMMARY:
Prospective, Open Label, Cohort Study in Traumatic Brain Injury Patients. The goal of this study is to assess the safety of NTx®-265. NTx®-265 will be administered over 9 days, and patients will be followed for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18-65
2. Written and informed consent from a legally acceptable representative
3. Moderate to severe traumatic brain injury (TBI) defined as Glasgow Coma motor (GCSm) score ≤5, post resuscitation.
4. Patient is <48hours from time of injury when the first dose of NTx™-265 is administered.
5. Reasonable expectation of availability to receive the full 9 day course of therapy and be available for follow up evaluations
6. Female patient is either:

   1. Not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral oophorectomy or hysterectomy) or
   2. If of childbearing potential, would agree to use two of the following reliable methods of birth control throughout the study, including the follow-up visits:

      * Condoms, sponge, foams, jellies, diaphragm or intrauterine device
      * A vasectomised partner
      * Abstinence
      * Note: Hormonal Based contraceptives are NOT permissible as one of the two forms of contraceptives for this study.

Exclusion Criteria:

1. Women who have been tested positive for pregnancy, or are breast-feeding or are not using a highly effective method of birth control that can be maintained for the duration of the study.
2. Bilaterally fixed pupils
3. Serum hemoglobin >160g/L (males) or >140g/L (female); or platelet count > 400,000/mm3
4. Advanced cardiac, pulmonary, hepatic or liver disease; the former will be operationally defined using NCI Toxicity Criteria (Grade 2 or higher).
5. Suspected anoxic or ischemic brain injury
6. Known endocrine or germ cell tumor
7. Serum billirubin > 1.5 x upper limit of normal (ULN).
8. Alkaline Phosphatase > 2.5 x ULN
9. AST and/or ALT > 2.5 x ULN
10. Creatinine > 2.0 x ULN
11. Patients with known or documented transferrin saturation < 20% or ferritin < 100ng/mL.
12. Male patients with known and documented elevated PSA levels, or a PSA level of ≥4ng/mL at screening.
13. Patients with known history or hypercoagulability, including known cardiolipin/antiphospholipid antibody syndrome.
14. Allergy or other contraindication to hCG including:

    1. Prior hypersensitivity to hCG preparations or one of their excipients.
    2. Primary ovarian failure.
    3. Uncontrolled thyroid or adrenal dysfunction.
    4. An uncontrolled organic intracranial lesion such as a pituitary tumor.
    5. Abnormal uterine bleeding of undetermined origin.
    6. Ovarian cyst or ovarian enlargement of undetermined origin.
    7. Sex hormone dependent tumors of the reproductive organs, accessory sex glands, and breasts.
15. Allergy or other contraindication to epoetin alfa:

    1. Who developed pure red cell aplasia following treatment with any erythropoiesis regulating hormones.
    2. With uncontrolled hypertension
    3. With known hypersensitivity to mammalian cell-derived products, albumin (human) or any component of the product
    4. Who for any reason cannot receive adequate antithrombotic treatment
16. A known diagnosis of cancer (except basal cell cancer).
17. Uncontrolled hypertension, defined as blood pressure persistently above 220 mm Hg systolic or 120 mm Hg diastolic despite antihypertensive therapy.
18. Use of either hCG or epoetin alfa within the previous 90 days.
19. Any condition known to elevate hCG, active in the prior 24 months e.g., choriocarcinoma or germ cell tumor.
20. Any patients living in a nursing home or supervised living center. Patients must be historically fully independent in all activities of daily living including banking, shopping, cooking, toileting, showering and dressing.
21. Any other medical condition, in the investigator's opinion, the patient should not be included in the trial.
22. Patients who cannot take anti-platelet or anti-coagulant therapy.
23. Pre-existing and active major psychiatric or other chronic Neurological disease.
24. Patients who have a history of substance abuse or dependency within 12 months prior to the study.
25. Currently participating in another investigational study
26. Polytrauma defined as an Abbreviated Injury Severity Score >3 in any area other than head.
27. Patients with evidence of an active or previous thrombotic event.
28. Patients with contraindications to MRI scans
29. Patients who are currently taking hormonal based contraceptives or hormonal replacement therapy in the past three (3) months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 months
  The primary endpoint for this study is safety. The following safety endpoints will be assessed:
  * Type, incidence, severity, timing, seriousness, and relatedness of adverse events.
  * Lower extremity deep vein ultrasound will be performed to identify and localize deep or superficial venous thrombosis.
  * Vital signs
  * Laboratory assessments. Particular attention will be paid to serial hemoglobin and hematocrit measurements.
  * DVT, PE, thromboembolism, MI and stroke.

SECONDARY OUTCOMES:
Efficacy | 6 months
  The following secondary endpoints will also be assessed in order to measure various aspects of neurological status:
  * GOSE at hospital discharge, 3, and 6 months post-TBI
  * Neurobehavioral Rating Score at hospital discharge, 3, and 6 months post TBI
  * Disability Rating Score at hospital discharge, 3, and 6 months post TBI

CONTACTS AND LOCATIONS:
Overall Officials: David A Zygun, MD, MSc, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Center, Calgary, Alberta, Canada